CLINICAL TRIAL: NCT00240838
Title: A Randomized, Double-Blind Study Evaluating Acetaminophen Extended Release Caplets (3900 mg/Day) and Ibuprofen (1200 mg/Day) in the Treatment of Post-Race Muscle Soreness.
Brief Title: An Effectiveness and Safety Study Comparing Acetaminophen (3900 mg/Day) to Ibuprofen (1200 mg/Day) in the Treatment of Post-Race Muscle Soreness.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002866
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Pain
Keywords: muscle soreness; pain, acetaminophen; ibuprofen
MeSH Terms: conditions — Pain; Myalgia

INTERVENTIONS:
Drug: acetaminophen extended release caplets

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of acetaminophen extended release caplets and ibuprofen in relieving the muscle soreness that occurs after a marathon.

DETAILED DESCRIPTION:
The objective of this randomized, double-blind study is to compare the effectiveness and safety of acetaminophen extended release caplets and ibuprofen in relieving the muscle soreness that occurs in subjects who complete a marathon. Subjects are randomized to receive acetaminophen extended release caplets, 3900 mg/day (two 650 mg caplets taken three times a day, for five days) or ibuprofen caplets, 1200 mg/day (two 200 mg caplets taken three times a day, for five days). The primary measurement of efficacy is the average change in muscle soreness from baseline for both the morning and evening assessments. Safety assessments consist of monitoring adverse events, and a physical examination including vital signs, weight, a review of concomitant medications, and a urine pregnancy test for female subjects. Two hypotheses are examined in a step-down approach. The first hypothesis is that acetaminophen extended release is not inferior to ibuprofen in relieving the muscle soreness that occurs after a marathon. If acetaminophen extended release is not inferior to ibuprofen in relieving the muscle soreness that occurs after a marathon, the second hypothesis is that acetaminophen extended release (3900 mg/day) is superior to ibuprofen (1200 mg/day) in relieving the muscle soreness that occurs after a marathon. Two acetaminophen 650 mg extended release caplets, taken by mouth, three times a day for five days or two ibuprofen 200 mg caplets, taken by mouth, three times a day for five days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must complete the marathon
* be able to swallow the study medication
* comply with study requirements regarding the use of any other pain medications before, during or after the marathon
* rate their muscle soreness on the evening after the marathon as at least a 4, on a zero-to-ten point scale
* if female, must not be pregnant or breastfeeding, and must be using an acceptable form of contraception

Exclusion Criteria:

* Previous diagnosis of osteoarthritis requiring pain medication therapy
* currently have a major medical illness
* have a history of cardiovascular disease, heat injury (heat exhaustion or heat stroke) or collapse during a running or endurance event
* known hypersensitivity to acetaminophen or ibuprofen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2003-05; Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Average change in muscle soreness from baseline for both morning and evening assessments.

SECONDARY OUTCOMES:
Average change in muscle soreness from baseline for morning assessments; Average change in muscle soreness from baseline for evening assessments; Average ratings of interference with 1) sleep; 2) morning activity; 3) ability to go for a run

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- See also: An Effectiveness and Safety Study comparing Acetaminophen (3900 mg/day) to Ibuprofen (1200 mg/day) in the Treatment of Post-Race Muscle Soreness. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=912&filename=CR002866_CSR.pdf